CLINICAL TRIAL: NCT05720156
Title: ImmuNomodulatory EffectS of PCSK9 Inhibition: A TaRgeted Molecular Imaging AppRoach
Brief Title: Immunomodulatory Effects of PCSK9 Inhibition
Acronym: INSPIRAR
Status: Withdrawn | Type: Observational
Why Stopped: Lack of Feasibility
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Mabel Toribio, Assistant Professor, Massachusetts General Hospital
Other Study IDs: 2022P002214
Record Dates: First submitted 2023-01-20; First posted 2023-02-09 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Atherosclerotic Cardiovascular Disease; Cardiovascular Diseases; Atherosclerosis; Arterial Inflammation; Vascular Diseases; Vascular Disease, Peripheral; Vascular Calcification; High Cholesterol/Hyperlipidemia; Heart Diseases; Heart Attack; Stroke; Cerebrovascular Accident; Carotid Artery Diseases; Carotid Atherosclerosis; Transient Ischemic Attack
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Arteritis; Vascular Diseases; Peripheral Vascular Diseases; Vascular Calcification; Hypercholesterolemia; Hyperlipidemias; Heart Diseases; Myocardial Infarction; Stroke; Carotid Artery Diseases; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: History of ASCVD, on high-intensity statins and initiating PCSK9 inhibitor therapy: History of ASCVD, on high-intensity statins and initiating PCSK9 inhibitor therapy
  Interventions: Other: 99mTc-tilmanocept SPECT/CT scanning
- Control group: No history of ASCVD, not on statins or initiating PCSK9 inhibitor therapy: No history of ASCVD, not currently on high-intensity statins, other lipid lowering therapy or initiating PCSK9 inhibitor therapy
  Interventions: Other: 99mTc-tilmanocept SPECT/CT scanning

INTERVENTIONS:
Other: 99mTc-tilmanocept SPECT/CT scanning — 99mTc-Tilmanocept SPECT/CT allows for visualization of macrophage-specific arterial infiltration

SUMMARY:
Cardiovascular disease (CVD) represents the leading cause of death worldwide. While medications, such as statins, significantly reduce atherosclerotic CVD (ASCVD) risk by lowering low density lipoprotein levels, they may also have pleiotropic effects on inflammation. The immunomodulatory effects of these medications are relevant to ASCVD risk reduction given that inflammation plays a central role in atherosclerotic plaque formation (atherogenesis) and influences the development of vulnerable plaque morphology. Patients on statins, however, may have residual inflammation contributing to incident ASCVD despite the potent LDL-lowering effects of statins. While new therapies, such as proprotein convertase subtilisin/kexin type 9 (PSCK9) inhibitors, further reduce incident ASCVD and drastically reduce LDL-C below that achieved by statin therapy alone, PCSK9 inhibitors may also have pleiotropic effects on inflammation. Thus, PCSK9 inhibitors may help reduce arterial inflammation to a level closer to that of patients without ASCVD. This study will apply a novel targeted molecular imaging approach, technetium 99m (99mTc)-tilmanocept SPECT/CT, to determine if residual macrophage-specific arterial inflammation is present with statin therapy and the immunomodulatory effects of PSCK9 inhibition. Given the continued high mortality and morbidity attributable to ASCVD, strong imperatives exist to better understand the immunomodulatory effects of lipid lowering therapies and residual inflammatory risk. This understanding, in turn, will inform the development of new ASCVD preventative and treatment strategies as well as elucidate other indications for established therapies.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 85 years of age
* CASE PARTICIPANTS ONLY: History of ASCVD (including a history of coronary artery disease, carotid artery disease, peripheral artery disease, acute coronary syndrome, percutaneous coronary intervention, coronary bypass surgery, carotid endarterectomy, stroke or TIA)
* CASE PARTICIPANTS ONLY: High-intensity statin therapy for at least 6 months prior enrollment and without an interruption of >1 month
* CASE PARTICIPANTS ONLY: Initiation of PCSK9 inhibition with either evolocumab or alirocumab (and not inclisiran - PSCK9 inhibition through small interfering RNA)

Exclusion Criteria:

* pregnancy or breastfeeding
* CONTROL PARTICIPANTS ONLY: No known history of ASCVD (including a history of coronary artery disease, carotid artery disease, peripheral artery disease, acute coronary syndrome, percutaneous coronary intervention, coronary bypass surgery, carotid endarterectomy, stroke or TIA)
* current treatment with prescription, systemic (oral, IV, IM or intra-articular) steroids or anti-inflammatory/immune suppressant medical therapies (excluding topical therapies, UV therapy, ASA-derivative therapies, or NSAIDS) for autoimmune/inflammatory diseases (psoriasis, RA, IBD, lupus), post-transplant care, asthma, or pain syndromes
* use of oral steroids or prescription oral anti-inflammatory/immune suppressant medication for > 7 days within the past 1 month
* use of IV, IM or intra-articular steroids or IV, IM or intra-articular anti-inflammatory/immune suppressant medication within the past 3 months
* Any prior use of PCSK9 inhibitors including both monoclonal antibodies or small interfering RNA
* CONTROL PARTICIPANTS ONLY: use of cholesterol lowering therapy (including statins, ezetimibe, bempedoic acid, PCSK9 inhibitors including both monoclonal antibodies or small interfering RNA, niacin, fibrates) or other lipid lowering agents associated with ASCVD risk reduction such as Vascepa. Cholesterol lowering therapies that that predominantly target triglycerides including over the counter omega-3 fatty acids and Lovaza are permitted.
* known allergy to dextrans and/or DTPA and/or radiometals
* significant radiation exposure (>2 CT angiograms) received within the past 12 months
* concurrent enrollment in another research study judged by the study investigators to interfere with the current study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Case: People with known ASCVD, on high-intensity statin therapy for at least 6 months and about to initiate PCSK9 inhibitor therapy
  Control: Healthy controls with no known ASCVD and not on statin
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-04-04 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Between-group difference (case participants versus control participants) in percent volume with aortic 99mTc-tilmanocept uptake across different uptake thresholds | Baseline
Change in the percent volume with aortic 99mTc-tilmanocept uptake across different uptake thresholds after PCSK9 inhibitor therapy for 12 months (case participants only) | Baseline and 12 Months

SECONDARY OUTCOMES:
Relationship between baseline immune cell subpopulations (cells/µL) and aortic volume with 99mTc-tilmanocept uptake | Baseline and 12 Months
Relationship between baseline markers of immune activation/ systemic inflammation and aortic volume with 99mTc-tilmanocept uptake | Baseline and 12 Months
Relationship between change in macrophage-specific arterial infiltration with PCSK9 inhibitors and change in immune cell subpopulations (cells/µL) | Baseline and 12 Months
Relationship between change in macrophage-specific arterial infiltration with PCSK9 inhibitors and change in markers of immune activation/ systemic inflammation | Baseline and 12 Months
Relationship between change in macrophage-specific arterial infiltration with PCSK9 inhibitors and baseline immune cell subpopulations (cells/µL) | Baseline and 12 Months
Relationship between change in macrophage-specific arterial infiltration with PCSK9 inhibitors and baseline markers of immune activation/ systemic inflammation | Baseline and 12 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No